CLINICAL TRIAL: NCT02805946
Title: Pharmacokinetics of Posaconazole (Noxafil®) as Prophylaxis for Invasive Fungal Infections
Acronym: PIRAÑA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UMCN-AKF16.01; 2016-001182-87 (EudraCT Number)
Record Dates: First submitted 2016-06-01; First posted 2016-06-20 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Allogeneic Stem Cell Transplant; Acute Graft Versus Host Disease; Acute Myeloid Leucaemia; Myelo Dysplastic Syndrome
MeSH Terms: interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intravenous followed by oral (Other): * Start with posaconazole IV 300mg BID on the first day. Posaconazole will be infused over a period of 90 minutes.
  * Days 2-7 patients will receive posaconazole IV 300mg QD.
  * Days 8-12 patients will receive posaconazole PO 300mg QD.
  * Days 13-16 patients will receive posaconazole PO 200mg QD.
  * 3 PK curves will be determined on days 7, 12 and 16 (after the 7th, 12th and 16th dosage).
  Interventions: Drug: posaconazole
- oral followed by intravenous (Other): * Start with posaconazole PO 300mg BID on the first day.
  * Days 2-7: patients will receive posaconazole PO 300mg QD.
  * Days 8-12: patients will receive posaconazole IV 300mg QD. Posaconazole will be infused over a period of 90 minutes.
  * Days 13-16 patients will receive posaconazole IV 200mg QD.
  * 3 PK curves will be determined on days 7, 12 and 16 (after the 7th, 12th and 16th dosage).
  Interventions: Drug: posaconazole

INTERVENTIONS:
Drug: posaconazole — iv versus oral
  Other Names: Noxafil

SUMMARY:
This study evaluates the the pharmacokinetics of posaconazole (new solid oral and IV) given as prophylaxis to patients who are at risk for developing fungal infections after receiving conditioning therapy (except strictly non-myeloablative (NMA)) for allogeneic Stem Cell Transplant (SCT), remission induction chemotherapy for acute myeloid leukemia (AML) or myelo dysplastic syndrome (MDS) or being treated for severe graft versus host disease (GvHD) and determines the impact of mucositis on the pharmacokinetics of posaconazole new solid oral.

DETAILED DESCRIPTION:
In 2014, the new intravenous and solid oral formulation of posaconazole were marketed. This offers new treatment possibilities, specifically in patients previously unable to attain adequate exposure to posaconazole solution. To the opinion of the researchers, only limited data are available on the pharmacokinetics (PK) of the new formulations of posaconazole, however, these use strictly selected patients or healthy volunteers, but more importantly, specific aspects related to the PK remain unsolved. Despite the fact that adequate exposure is attained using the new solid oral formulation, it is hypothesized that oral bioavailability of posaconazole may be impacted during mucositis. Whether mucosal barrier injury impacts the absorption of posaconazole or alters presystemic clearance is still unknown. Therefore, it seems prudent to conduct a trial in a group of patients that will experience a severe degree of mucositis to identify changes in absorption of posaconazole and resolving the impact of various stages of mucositis on the PK of posaconazole by linking PK of posaconazole to markers of mucositis (citrulline). This research may also serve as a model for other drugs and allows for direct translations in improving patient care. For this purpose it is needed to determine the PK using both IV and PO dosing of posaconazole.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
2. Subject is at least 18 years of age on the day of providing informed consent.
3. Patient receives immunosuppressive therapy for acute or chronic GVHD grade II-IV, reduced intensity conditioning regimens for allogeneic stem cell transplant, or first remission induction chemotherapy for AML/MDS.
4. In case of acute GVHD grade II-IV, patient has received less than 1 week of immunosuppressive therapy.
5. If a woman, is neither pregnant nor able to become pregnant and is not nursing an infant.
6. Has an ALAT <200U/L, ALAT <225U/L, alkaline phosphatase <60 U/L and a bilirubin level <50 μmol/L.
7. Subject is capable of receiving oral tablets.
8. Subject is managed with a central venous or arterial catheter.

Exclusion Criteria:

1. Documented history of sensitivity to medicinal products or excipients similar to those found in the posaconazole preparation.
2. Relevant history or presence of cardiovascular disorders (specifically QTc-time prolongation).
3. Inability to understand the nature of the trial and the procedures required
4. Any signs or symptoms of invasive fungal disease or the use of antifungal drugs within the previous month.
5. Has previously participated in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-09-07 (Actual)

PRIMARY OUTCOMES:
exposure to posaconazole (Area Under the Curve) when administered intravenously and orally (tablet formulation) | day 7, day 12 and day 16
  Plasma samples drawn on t=0 (pre-dose), 0.5, 1 (just prior to end of infusion), 2, 3, 4, 6, 8, 10, 12, 18 and 24 hours post infusion or post intake will be taken op day 7, day 12 and day 16 to determine posaconazole concentrations. Area Under the Curve of two routes of administration and two dosing regimens will be determined.
impact of mucositis (determined by citrulline concentrations) on exposure (AUC) to posaconazole. | day 7, day 12 and day 16
  Full pharmacokinetic curve (plasma samples drawn on t=0 (pre-dose), 0.5, 1 (just prior to end of infusion), 2, 3, 4, 6, 8, 10, 12, 18 and 24 hours post infusion or post intake) will be taken op day 7, day 12 and day 16 (posaconazole). Impact of mucositis on oral absorption will be determined by comparing AUCs after intravenous administration with oral (tablet) administration in patients with mucositis.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Brüggemann, PhD, PharmD, Principal Investigator — Radboud University Medical Center
Locations (2):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No